CLINICAL TRIAL: NCT05108402
Title: Comparative Evaluation on Blood Pressure Effect of an Equivalent Sodium Intake, in the Form of Bicarbonate or Chloride, for Hypertensive Subjects.
Brief Title: Comparison on Blood Pressure Effect of an Equivalent Sodium Intake, With Different Nature, for Hypertensive Subjects
Acronym: SODIVASC-II
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: RBHP 2021 PICKERING 3; 2021-A01134-37 (Other: ANSM)
Record Dates: First submitted 2021-09-09; First posted 2021-11-04 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-09

CONDITIONS: Hypertension
Keywords: Sodium intake; Blood pressure; high blood pressure; bicarbonate sodium; chloride sodium; NaCl sensitive
MeSH Terms: conditions — Hypertension | interventions — Immunophenotyping

STUDY DESIGN:
Intervention Model Description: Single-center, randomized study, organized in 2 stages.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Bottle of water (Experimental): After inclusion in the study, the patients are phenotyped between V1 and V4. Following this, they will be separated into 2 groups: "NaCl sensitive" patients and "non-NaCl sensitive" patients. The non-sensitive group will drop out of the study, while the others will be randomized to one of the 2 treatment arms: bottle of water or sachet of salt.
  Interventions: Diagnostic Test: Phenotyping; Dietary Supplement: Drug intake
- Salt sachet (Active Comparator): After inclusion in the study, the patients are phenotyped between V1 and V4. Following this, they will be separated into 2 groups: "NaCl sensitive" patients and "non-NaCl sensitive" patients. The non-sensitive group will drop out of the study, while the others will be randomized to one of the 2 treatment arms: bottle of water or sachet of salt.
  Interventions: Diagnostic Test: Phenotyping; Dietary Supplement: Drug intake
- No treatment (Other): After inclusion in the study, the patients are phenotyped between V1 and V4. Following this, they will be separated into 2 groups: "NaCl sensitive" patients and "non-NaCl sensitive" patients. The non-sensitive group will drop out of the study, while the others will be randomized to one of the 2 treatment arms: bottle of water or sachet of salt.
  Interventions: Diagnostic Test: Phenotyping

INTERVENTIONS:
Diagnostic Test: Phenotyping — After inclusion in the study, between V1 and V4, patients will be phenotyped among: "NaCl sensitive" patients and "non-NaCl sensitive" patients. they will have a low sodium diet for 2 weeks. The first week without salt supplementation and the second with salt supplementation. At the end of V4, if patient is "NaCl sensitive" he will continue into treatment period and go through randomization, and for patient "non-NaCl sensitive" they will drop out of study.
Dietary Supplement: Drug intake — After being phenotyped, "NaCl sensitive" patients will continue the study in one of the 2 treatments arms : royal water (bottle) or salt sachet.
  Arms: Bottle of water; Salt sachet

SUMMARY:
Numerous large-scale epidemiological studies have made it possible to establish a link between the average consumption of table salt (sodium chloride) and blood pressure figures. In France, according to the French Agency for Food, Environmental and Occupational Health & Safety (ANSES), salt intakes could be estimated from 2 national food consumption surveys INCA 1 and INCA 2. This made it possible to take a photograph of food consumption habits and to show that the average consumption of salt contained in food in France is 8.7g/day for men and 6.7g/day for women. To these contributions must also be added 1 to 2g of salt for the resalting and the cooking water. According to the food consumption survey INCA 3, french plate still contains a large part of processed foods and still a little too much salt (on average 9g/day for men and 7g/day for women at compare with the objectives of the National Health Nutrition Program of 8g/day and 6.5g/day respectively). In addition, the World Health Organization (WHO) recommends consuming less than 5g of salt per day.

In this context, sodium intake through mineral water was also questioned. Both in terms of basic and clinical research, the biological effects of dietary sodium chloride intake have been the subject of a great deal of work for several decades. The mechanisms of transmission in the induced or hemodynamic effects related to the absorption of Na multiple debates and their impact on cardiovascular risks remain very uncertain. Work has shown that all subjects do not react homogeneously to sodium chloride intakes, thus determining what are called "NaCl-sensitive" people who in a situation of major sodium intake will show an increase of peripheral vascular resistance and an increase in blood pressure, much more marked than in subjects called " NaCl resistant ".

"NaCl-sensitive" people represent 10 to 30% of the population, with notable differences according to ethnic origins, regions and continents. A marked overrepresentation of this phenotype is observed in patients with hypertension or with a family history of hypertension.

Furthermore, studies conducted on animals and humans show that sodium intake does not have the same impact on the parameters mentioned above, depending on whether it is in the form of chloride or bicarbonate salt.

On the basis of these elements, the investigators developed a clinical study protocol intended to demonstrate a possible differential effect in the biological effects of the same sodium orally intake (2.56g per day), depending on the salt origin.

DETAILED DESCRIPTION:
This single-center, randomized study, aim to determine the difference in absorption between sodium depending on its nature: bicarbonate (NaHCO3) or chloride (NaCl), and the effect of those types of sodium on blood pressure.

In order to realize it, 206 volunteers will be include to assess whether or not they are a "NaCl sensitive volunteer" phenotype.

The study will be carried out on 34 of NaCl sensitive volunteer which will take the sodium dietary supplements. The 2 dietary supplements are table salt (sachet) or bottled water. They will be test in a cross-over design during 2 periods of 1 week separated from 1 week of a washing-out period.

The primary objective will be to compare mean arterial pressure (MAP) resulting from daily supplementation of 2.56 g of sodium (111 mmol), in addition to the food intake of a low-sodium diet from V2 to the end of the study (<5g of NaCl / day), for 7 days, either as sodium chloride or as sodium bicarbonate in hypertensive subjects.

This clinical trial will be separated in 2 phases:

1. Phenotyping (4 visits): to determine if the volunteer is "NaCl sensitive volunteer" or not

   1. V1 (day -28/D-28) = inclusion and beginning of phenotyping phase,
   2. V2 (day -21/D-21) = start of a low-sodium diet (<5g of NaCl / day),
   3. V3 (day -14/D-14) = daily supplementation of sodium chloride for 7 days (9.78g/day),
   4. V4 (day -7/D-7) = "NaCl sensitive volunteer" assessment, end of study for "NaCl non-senstive volunteers".
2. Treatment period for "NaCl sensitive volunteer" with dietary supplement intake in a cross-over design:

   1. PC1 (day 0/D0) = beginning of treatment period 1,
   2. PC2 (day 3/D3) = volunteer contact to make sure he is all right,
   3. V5 (day 7/D7) = end treatment period 1,
   4. PC3 (day 14/D14) = beginning of treatment period 2,
   5. PC4 (day 17/D17) = volunteer contact to make sure he is all right,
   6. V6 (day 21/D21) = end of treatment period 2 and of the study.

The protocol includes a total of 6 visits to PIC/CIC Inserm 1405 of the Clermont-Ferrand University Hospital.

The maximum duration of the study will be of 7 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Systolic blood pressure between 135-160 mmHg and diastolic 85-100 in self-measurement, untreated or treated but not balanced under treatment,
* Father or mother hypertensive,
* Weight ≥ 50 kg
* Absence of known heart disease,
* Brachialis perimeter between 22 and 42 cm,
* Creatinine clearance within the standards dating from less than 12 months, (GFR> 60ml / min / 1.73m²),
* Agreeing to drink sparkling water during one of the study periods,
* Effective contraception for female subjects of childbearing age,
* Cooperation and understanding sufficient to comply with the requirements of the test,
* Affiliated with a Social Security scheme,
* Agreeing to give written consent,
* Registration or acceptance of registration in the national register of volunteers participating in research.

Exclusion Criteria:

* Consumption of more than 5g/day of salt in the protocol diet (evaluated by natriuresis analyzed in V3)
* Systemic corticosteroid therapy
* Taking prohibited drugs (see list) and at the judgment of the investigator.
* Suffering from pulmonary hypertension
* Woman of childbearing age not using an effective contraceptive method, pregnant or breastfeeding woman,
* History of cardiomyopathy or ischemic heart disease,
* Absence of sinus rhythm,
* Renal failure (DFG <60 ml/min/1.73m²),
* Comorbidity incompatible with the study,
* BMI> 35 kg/m2,
* Disabling cognitive disorders,
* Anxiety when taking measurements alone at home at the judgment of the investigator,
* Diabetes (Type I and II)
* Chronic alcoholism,
* Sports activity deemed to be intense (more than 3 hours / week of intense sport),
* Extreme sweating activity (Sauna, Hammam),
* During participation in another clinical trial, or in the exclusion period, or having received a total amount of compensation greater than 4,500 euros over the 12 months preceding the start of the trial,
* Benefiting from a legal protection measure (curatorship, guardianship, deprived of freedoms, safeguard of justice)
* Not affiliated with the French Social Security scheme.
* Any history deemed significant by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Change from mean blood pressure (MBP) at Day 21 | Day 21
  Comparison between blood pressure data recorded by the volunteer between the 2 weeks of treatment (measurement during 2 days before Day 7 and 2 days before Day 21).
  Recording of systolic and diastolic blood pressure will be made by the patient at home with the Microlife BP A200 device, in the morning and evening.
  Comparison of the data collected from these 2 weeks of treatment will allow us to meet the main objective of the study.

SECONDARY OUTCOMES:
Change from mean blood pressure (MBP) at Day -7 | Day -7
  Comparison between blood pressure data recorded by the volunteer for the last 2 days before Day -14 and the last 2 days before Day -7.
  Recording of systolic and diastolic blood pressure will be made by the patient at home with the Microlife BP A200 device, in the morning and evening to determine if the subject is "NaCl sensitive" or not.
Weight | Day -28, Day -21, Day -14, Day -7, Day 7 and Day 21
  Measure of patient weight (in kilograms) using a weighing machine.
Body composition analysis | Day -21, Day -14, Day -7, Day 7 and Day 21
  Measurement of water quantities in the body, fat and muscle, will be analyzed using an non-invasive device by impedance measurement. Patient will be comfortably installed in a quiet room, lying down on a bed where two electrodes will be applied, one at the level of the hand, the other at the level of the foot.
Optional genotyping | One time at Day -28
  With patient agreement: 1 tube of blood (9mL) used for genetics analysis: genotyping
Plasma renin dosage on fasted state | Day -28, Day -14, Day -7, Day 7 and Day 21
  Concentration of renin in plasma (ng/mL/h) will be measured on fasted state.
Plasma Angiotensin II dosage on fasted state | Day -28, Day -14, Day -7, Day 7 and Day 21
  Concentration of angiotensin II (µg/L) in plasma will be measured on fasted state.
Plasma Aldosterone dosage on fasted state | Day -28, Day -14, Day -7, Day 7 and Day 21
  Concentration of aldosterone (pg/mL) in plasma will be measured on fasted state.
Plasma potassium dosage on fasted state | Day -28, Day -14, Day -7, Day 7 and Day 21
  Concentration of potassium (mmol/L) in plasma will be measured on fasted state.
Plasma sodium dosage on fasted state | Day -28, Day -14, Day -7, Day 7 and Day 21
  Concentration of sodium (mmol/L) in plasma will be measured on fasted state.
Plasma calcium dosage on fasted state | Day -28, Day -14, Day -7, Day 7 and Day 21
  Concentration of calcium (mmol/L) in plasma will be measured on fasted state.
Plasma chlorine dosage on fasted state | Day -28, Day -14, Day -7, Day 7 and Day 21
  Concentration of chlorine (mmol/L) in plasma will be measured on fasted state.
Plasma protein dosage on fasted state | Day -28, Day -14, Day -7, Day 7 and Day 21
  Concentration of protein (mmol/L) in plasma will be measured on fasted state.
Serum creatinine dosage on fasted state | Day -28, Day -14, Day -7, Day 7 and Day 21
  Concentration of creatinine (mmol/L) in serum will be measured on fasted state.
Serum urea dosage on fasted state | Day -28, Day -14, Day -7, Day 7 and Day 21
  Concentration of urea (mmol/L) in serum will be measured on fasted state.
Sodium concentration in 24h urine | Day -28, Day -14, Day -7, Day 7 and Day 21
  Concentration of sodium in urine (mmol/24h) will be measured.
Potassium concentration in 24h urine | Day -28, Day -14, Day -7, Day 7 and Day 21
  Concentration of potassium in urine (mmol/24h) will be measured.
Creatinine concentration in 24h urine | Day -28, Day -14, Day -7, Day 7 and Day 21
  Concentration of creatinine in urine (mmol/24h) will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Gisele PICKERING, MD, Principal Investigator — Platform of Clinical Investigation/Clinical Investigation Center French Institute of Health and Medical Research-1405 63000 Clermont-Ferrand FRANCE
Locations (1):
- Platform of Clinical Investigation / Clinical Investigation Center French Institute of Health and Medical Research-1405 University Hospital, Clermont-Ferrand, Auvergne, France

REFERENCES:
- See also: Clinical trial link for previous clinical trial on the same subject — https://clinicaltrials.gov/ct2/show/NCT02561325?term=sodivasc&draw=2&rank=1